CLINICAL TRIAL: NCT02348502
Title: Sustained Viral Response and HBsAg Level Changes in Chronic Hepatitis B Patients Who Achieved HBsAg Level≤100 IU/ml After Completed Interferon Therapy
Brief Title: Sustained Viral Response in Patients Achieved HBsAg Level≤100 IU/ml After Completed Interferon Treatment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Beijing Ditan Hospital (Other)
Responsible Party: Principal Investigator, Yao Xie, liver diseases center, Beijing Ditan Hospital
Other Study IDs: DTXY003
Record Dates: First submitted 2015-01-22; First posted 2015-01-28 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Hepatitis B
Keywords: HBsAg loss; interferon; HBV reaction; Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Chronic hepatitis B (CHB) is a serious liver disease worldwide, and the leading cause of cirrhosis and hepatocellular carcinoma (HCC). HBsAg loss/seroconversion is considered to be the ideal endpoint of antiviral therapy in both HBeAg-positive and -negative patients, and the ultimate treatment goal in CHB, However HBsAg loss occurred rarely by interferon treatment. Although It was reported that in nature history HBsAg level≤100 IU/ml can bring good long term outcomes in patients with chronic hepatitis B. it was not clear whether patients who achieved HBsAg level≤100 IU/ml by interferon treatment could maintain sustained viral response and the state of HBsAg level≤100 IU/ml.

DETAILED DESCRIPTION:
The patients with chronic hepatitis B and achieved HBsAg level≤100 IU/ml after completed interferon treatment will be enrolled and observed for 96 weeks. Serum HBV DNA, HBsAg, anti-HBs, HBeAg, and anti-HBe will be measured every 3 months during the observation period, liver function tests were performed every 3 months also. The liver ultrasonic examination would be taken every 3-6 months. The primary endpoint is HBV DNA reaction. The secondary endpoints is HBsAg loss.

ELIGIBILITY:
Inclusion Criteria:

* patients who had chronic hepatitis B and achieved HBsAg level≤100 IU/ml with undetectable HBV DNA level by interferon treatment

Exclusion Criteria:

* Active consumption of alcohol and/or drugs
* Co-infection with human immunodeficiency virus, hepatitis C virus, or hepatitis D virus
* History of autoimmune hepatitis
* Psychiatric disease
* Evidence of neoplastic diseases of the liver

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: the study population in this study were composed of patients who had chronic hepatitis B and achieved HBsAg level≤100 IU/ml with undetectable HBV DNA level after interferon treatment, and serum HBsAg and HBV DNA would be tested every 3 months for 96 weeks after finished treatment. Sustained viral response defined as serum HBV DNA maintaining undetectable during the observation period. HBsAg loss is defined as HBsAg level reached the value lower than the low limited value.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2013-01; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
the rate of sustained viral response | 96 weeks
  The serum HBV DNA will be tested every 3 month for 96 weeks after completed treatment in chronic hepatitis B patients who achieved serum HBsAg level≤100 IU/ml with HBV DNA undetectable by interferon therapy. The rate of sustained viral response defined HBV DNA level maintaining undetectable during observation period will be evaluated, and HBV reaction is defined as serum HBV DNA reverse back to detectable level.

SECONDARY OUTCOMES:
the rate of HBsAg loss | 96 weeks
  The serum HBsAg level will be tested every 3 month after completed treatment. The rate of HBsAg loss defined as HBsAg level reached the value lower than the low limited value will be evaluated after 96 weeks follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- liver disease center, Beijing Ditan Hospital, Beijing, Beijing Municipality, China